CLINICAL TRIAL: NCT01079988
Title: A Phase IV Open Label, Multicentre, Investigational Study of the Therapeutic Options for Subjects Discontinuing Efalizumab Therapy and Experiencing Inflammatory Disease Recurrence
Brief Title: Study of Therapeutic Options for Subjects Discontinuing Efalizumab and Experiencing Disease Recurrence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25180
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Results first posted 2010-05-11 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-01

CONDITIONS: Psoriasis
Keywords: Psoriasis; Discontinuation of efalizumab; Managing inflammatory recurrence
MeSH Terms: conditions — Psoriasis | interventions — Cyclosporins; Retinoids; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cyclosporin (Experimental): Starting dose 4.0 - 5.1 mg/kg/day until clinical improvement. Upon clinical improvement, cyclosporin dose to be tapered by 50% every two weeks.
  Interventions: Drug: Cyclosporins
- Retinoids (Experimental): Starting dose 25 - 50 mg/day until clinical improvement. Upon clinical improvement, retinoid dose to be reduced by 50%. Thereafter, treatment to be continued for 8 weeks and then stopped.
  Interventions: Drug: Retinoids
- Systemic corticosteroids (Experimental): Starting dose 0.25 - 0.5 mg/kg/day until clinical improvement. Upon clinical improvement, corticosteroid dose to be reduced by 50%. Thereafter, corticosteroids to be weaned by 50% every 2 weeks.
  Interventions: Drug: Systemic corticosteroids
- Methotrexate (Experimental): Starting dose 20 - 25 mg per week until clinical improvement. Upon clinical improvement, dose to be reduced by 25%. Thereafter, methotrexate dose to be reduced by 25% every two weeks.
  Interventions: Drug: Methotrexate
- Systemic corticosteroids/methotrexate (Experimental): Corticosteroid starting dose 0.25 - 0.5 mg/kg/day until clinical improvement. Upon clinical improvement, corticosteroid dose to be reduced by 50%.
  Thereafter, to be weaned by 50% every 2 weeks. Methotrexate starting dose 20 - 25 mg per week until clinical improvement. Upon clinical improvement, dose to be reduced by 25%. Thereafter, to be reduced by 25% every two weeks.
  Interventions: Drug: Systemic corticosteroids/methotrexate

INTERVENTIONS:
Drug: Cyclosporins — Starting dose 4.0 - 5.1 mg/kg/day until clinical improvement. Upon clinical improvement, cyclosporin dose to be tapered by 50% every two weeks.
  Arms: Cyclosporin
Drug: Retinoids — Starting dose 25 - 50 mg/day until clinical improvement. Upon clinical improvement, retinoid dose to be reduced by 50%. Thereafter, treatment to be continued for 8 weeks and then stopped.
  Arms: Retinoids
Drug: Systemic corticosteroids — Starting dose 0.25 - 0.5 mg/kg/day until clinical improvement. Upon clinical improvement, corticosteroid dose to be reduced by 50%. Thereafter, corticosteroids to be weaned by 50% every 2 weeks.
  Arms: Systemic corticosteroids
Drug: Methotrexate — Starting dose 20 - 25 mg per week until clinical improvement. Upon clinical improvement, dose to be reduced by 25%. Thereafter, methotrexate dose to be reduced by 25% every two weeks.
  Arms: Methotrexate
Drug: Systemic corticosteroids/methotrexate — Upon clinical improvement, corticosteroid dose to be reduced by 50%. Thereafter, to be weaned by 50% every 2 weeks. Methotrexate starting dose 20 - 25 mg per week until clinical improvement. Upon clinical improvement, dose to be reduced by 25%. Thereafter, to be reduced by 25% every two weeks.
  Arms: Systemic corticosteroids/methotrexate

SUMMARY:
This is a pilot investigational study of the appropriate therapeutic regimens to treat subjects experiencing inflammatory recurrence (rebound) of psoriatic disease upon discontinuation of efalizumab therapy and of the biological mechanisms involved in inflammatory disease recurrence and control.

ELIGIBILITY:
Inclusion Criteria:

* Participation in Genentech study ACD2601g, Genentech study HUPA 600 or Serono study IMP24011.
* Inflammatory psoriasis disease recurrence occurring up to 2 months after discontinuation of efalizumab that required immediate therapeutic control in the opinion of the Investigator. Psoriasis had to be rapidly developing, symptomatic and inflammatory in nature.
* Written informed consent, given prior to any study-related procedure not part of the subject's normal medical care, with the understanding that the subject could withdraw consent at any time without prejudice to his or her future medical care.
* Female subjects had to be neither pregnant nor breast-feeding, and had to lack childbearing potential, as defined by either:

  * Being post-menopausal or surgically sterile, or
  * Using an accepted form of contraception.
* Confirmation that the subject was not pregnant had to be established by a negative urinary hCG test at SD1. A pregnancy test was not required if the subject was post-menopausal or surgically sterile.
* Outpatient status at the time of enrolment.

Exclusion Criteria:

* Disease recurrence that was part of the natural disease progression, was not inflammatory in nature, and was not related to efalizumab study medication in the previous study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2004-02; Primary Completion 2004-12 (Actual); Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Natta, MD, Study Director — Merck Serono SA

REFERENCES:
- [Result] Papp KA, Toth D, Rosoph L, on behalf of the 25180 study group. Approaches to discontinuing efalizumab: results of an open-label study comparing different transitioning therapies. Abstract for presentation at EADV2005, Sofia, Bulgaria, 19-22 May 2005

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Initiation Date: 24 February 2004 (first patient, first visit) Study Completion Date: 21 December 2004 (last patient, last visit) Study Centres: 9 clinical centres in Canada
Pre-assignment Details: Subjects who satisfied the study's entry criteria were assigned to receive one of five treatment regimens involving accepted therapies for moderate to severe psoriasis
Period: Overall Study
Arm/Group | Cyclosporin | Retinoids | Systemic Corticosteroids | Methotrexate | Systemic Corticosteroids/Methotrexate
Started | 10 | 1 | 8 | 20 | 2
Completed | 9 | 1 | 8 | 17 | 1
Not Completed | 1 | 0 | 0 | 3 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyclosporin | Retinoids | Systemic Corticosteroids | Methotrexate | Systemic Corticosteroids/Methotrexate | Total
Number analyzed (Participants) | 10 | 1 | 8 | 20 | 2 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (12) | 41 | 44 (11) | 49 (10) | 47 (3) | 46 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 3 | 7 | 1 | 16
  Male | 5 | 1 | 5 | 13 | 1 | 25
Region of Enrollment [Number; unit: participants]
  Canada | 10 | 1 | 8 | 20 | 2 | 41

OUTCOME MEASURES:

1. Primary Outcome: Physician's Global Assessment (PGA) of Change Over Time (Good or Better)
Description: The PGA response was classified according to the following categories by changes in all clinical signs and symptoms as compared to baseline:
  Cleared: Remission except for residual manifestations such as mild erythema (100% improvement) Excellent: Improvement of 75%-99% except for residual manifestations such as mild erythema Good: Improvement of 50%-74%
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Cyclosporin | Retinoids | Systemic Corticosteroids | Methotrexate | Systemic Corticosteroids/Methotrexate
Number analyzed (Participants) | 10 | 1 | 8 | 20 | 2
participants | 7 | 0 | 2 | 9 | 0

2. Secondary Outcome: Patient's Global Psoriasis Assessment (PGPA)
Description: The PGPA consisted of a single self-explanatory item:
  On a scale from 0 to 10, with 0 being no psoriasis and 10 the worst psoriasis that you can imagine, please rate the state of your psoriasis right now.
  Note: Consider only your skin condition and do not consider other aspects that may be related to your psoriasis (such as psoriatic arthritis).
Time Frame: 12 weeks
Population: One patient withdrew
Measure: Mean (Standard Deviation); unit: PGPA score
Arm/Group | Cyclosporin | Retinoids | Systemic Corticosteroids | Methotrexate | Systemic Corticosteroids/Methotrexate
Number analyzed (Participants) | 10 | 1 | 8 | 19 | 2
PGPA score | 5.1 (2.4) | 4.0 | 5.5 (2.8) | 4.8 (2.7) | 4.5 (0.7)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored throughout the study
Description: Information about adverse events was obtained at study visits following physical examination, through spontaneous reports by the subjects and through questioning of the subjects. Adverse event data could also be obtained from subject diary cards, but such information had to be reviewed and assessed medically before it was transcribed to the CRF.
Arm/Group | Cyclosporin | Retinoids | Systemic Corticosteroids | Methotrexate | Systemic Corticosteroids/Methotrexate
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/1 | 0/8 | 0/20 | 0/2
Other Adverse Events (participants affected / at risk) | 9/10 | 0/1 | 4/8 | 11/20 | 0/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclosporin (N=10) | Retinoids (N=1) | Systemic Corticosteroids (N=8) | Methotrexate (N=20) | Systemic Corticosteroids/Methotrexate (N=2)
Influenza (Infections and infestations) | 1 | 0 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Herpes zoster ophthalmic (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Tongue disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 2 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0
Rigors (General disorders) | 0 | 0 | 1 | 0 | 0
Chronic obstructive airways disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other